CLINICAL TRIAL: NCT03352245
Title: Assessing the Feasibility of a Patient-centered Activity Regimen in Patients With Advanced Stage Lung Cancer
Brief Title: Feasibility of an Activity Regimen in Patients With Advanced Stage Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Medical University of South Carolina (Other); VA Connecticut Healthcare System (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000022225; 1P50CA196530-01 (NIH)
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Lung Neoplasm Malignant
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Prescribed Activity designed to improve patient participation and adherence to prescriptions to increase physical activity and will include: (1) an educational session at enrollment, (2) subject communication via tailored electronic messaging, and (3) a wrist-bound device (FitBit Flex 2).
  Interventions: Behavioral: Prescribed Activity
- Control Group (No Intervention): Usual care group will receive standard of care management from their Oncologist.

INTERVENTIONS:
Behavioral: Prescribed Activity — Educational session at enrollment, increase subject communication via tailored electronic messaging, and use of a wrist-bound device (FitBit Flex 2)
  Arms: Intervention Group

SUMMARY:
The investigators will evaluate the feasibility of implementing a low-intensity, patient-centered activity regimen (PCAR) that prioritizes education and communication over a 12-week period in advanced stage lung cancer patients. The primary outcomes will include number of patients increasing their overall step count over the study period and adherence to step count recommendations. Secondary outcomes will include quality of life (QoL), dyspnea, and depression scores before and after the intervention as well as a patient feedback questionnaire (to guide further interventions). The goals are to increase overall step count and obtain adherence of >50% of participants. The investigators will also assess whether the physical activity regimen influences markers of inflammation and glucose control and novel markers of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of advanced non-small cell stage lung cancer (NSCLC)
* Approval of the treating clinician
* Adult patients (age >21 years) willing to wear a FitBit® device (FitBit, Inc., San Francisco, CA)
* Access to a smartphone, agree to receive twice/daily text messages for 12 weeks (including any costs), and willingness to download the FitBit application to their smartphone.
* Low activity level as judged by a brief physical activity questionnaire (i.e., <150 minutes/week of moderate-intensity exercise, <75 minutes/week of vigorous aerobic exercise, or an equivalent combination).

Exclusion Criteria:

* Memory impairment (as judged by the treating clinician)
* Communication impairment (as judged by the treating clinician)
* Treating clinician's request not to alter physical activity
* Physical inability to safely walk (as judged by the treating clinician)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Bade, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bade BC, Gan G, Li F, Lu L, Tanoue L, Silvestri GA, Irwin ML. "Randomized trial of physical activity on quality of life and lung cancer biomarkers in patients with advanced stage lung cancer: a pilot study". BMC Cancer. 2021 Apr 1;21(1):352. doi: 10.1186/s12885-021-08084-0. PMID 33794808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.55 (7.28) | 63.20 (63.50) | 64.88 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 8 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 16 | 34
  Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Step Count
Description: Participants will wear a Fitbit wrist band that will record step count.
Time Frame: baseline to 12 weeks
Population: This outcome was measured only in the intervention group.
Measure: Mean (Full Range); unit: Steps
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 0
Steps
  Baseline | 4707 [1,568 to 12,222] |
  6 weeks | 5605 [1,079 to 9,764] |
  12 weeks | 4606 [746 to 10,238] |

2. Primary Outcome: Number of Weeks Participants Adhered to Step Count Recommendations
Description: Exercise Adherence will be defined as (the number of weeks a subject follows the activity prescription)/(the number of "usable" weeks). A week is considered "usable" if 5/7 days of step counts are available, and days with <200 steps/day are considered not usable.
Time Frame: baseline to 12 weeks.
Population: This outcome was measured only in the intervention group. The 19 participants were each followed for 12 weeks. Thus 19 participants were followed for a total of 228 weeks.
Measure: Count of Units; unit: Weeks
Units Other Than Participants: Weeks
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 0
Number analyzed (Weeks) | 228 | 0
Weeks | 47 |

3. Secondary Outcome: Dyspnea
Description: Assessed via self-report using the Modified Medical Research Council. Dyspnea Scale, a single-item scale scored 0-4; higher score indicates worse dyspnea.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
score on a scale | -0.04 (0.15) | -0.07 (0.15)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.889, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.20

4. Secondary Outcome: Depression
Description: Assessed via self-report using the Patient Health Questionnaire, Depression Module (PHQ-9). a 9-item questionnaire that assesses depressive symptoms over the preceding two weeks. Each item is scored 0-3 (0 = "Not at all"; 1 = "Several days"; 2 = "More than half of days"; 3 = "Nearly every day"). A total score is calculated by taking the sum of questions 1-9, and a higher score indicates worse depression.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
score on a scale | -0.83 (0.65) | 0.31 (0.68)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Net) = -1.14, Standard Error of Mean 0.88

5. Secondary Outcome: Change in Quality of Life: Global Health Status
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales:
  Global health status/Quality of Life (QoL) scale, range 0-100, higher score = better quality of life.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 3.16 (4.11) | -4.63 (4.20)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.166, Mixed Models Analysis; Mean Difference (Net) = 7.79, Standard Error of Mean 5.51

6. Secondary Outcome: Change in Quality of Life: Physical Functioning
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the 5 functional scales measure physical functioning.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 4.11 (2.50) | 4.74 (2.54)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.853, Mixed Models Analysis; Mean Difference (Net) = -0.64, Standard Error of Mean 3.41

7. Secondary Outcome: Change in Quality of Life: Role Functioning
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the 5 functional scales measures role functioning.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 8.09 (5.33) | -8.95 (5.45)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Net) = 17.04, Standard Error of Mean 7.16

8. Secondary Outcome: Change in Quality of Life: Emotional Functioning
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the 5 functional scales measures emotional functioning.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 2.68 (2.89) | 3.11 (2.95)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.911, Mixed Models Analysis; Mean Difference (Net) = -0.43, Standard Error of Mean 3.83

9. Secondary Outcome: Change in Quality of Life: Fatigue
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the symptom scale measures fatigue.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | -4.43 (4.85) | 0.75 (4.97)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.456, Mixed Models Analysis; Mean Difference (Net) = -5.18, Standard Error of Mean 6.88

10. Secondary Outcome: Change in Quality of Life: Cognitive Functioning
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the 5 functional scales measures cognitive functioning.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 0.41 (2.26) | 2.47 (2.31)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.515, Mixed Models Analysis; Mean Difference (Net) = -2.05, Standard Error of Mean 3.13

11. Secondary Outcome: Change in Quality of Life: Nausea/Vomiting
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the symptom scale measures nausea and vomiting The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | -2.44 (4.18) | 6.21 (4.28)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.144, Mixed Models Analysis; Mean Difference (Net) = -8.65, Standard Error of Mean 5.80

12. Secondary Outcome: Change in Quality of Life: Pain
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the symptom scale measures pain.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 1.67 (4.77) | 1.26 (4.87)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.948, Mixed Models Analysis; Mean Difference (Net) = 0.41, Standard Error of Mean 6.28

13. Secondary Outcome: Change in Quality of Life: Social Functioning
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the 5 functional scales measures social functioning.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | -4.22 (5.38) | 4.40 (5.50)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.254, Mixed Models Analysis; Mean Difference (Net) = -8.62, Standard Error of Mean 7.45

14. Secondary Outcome: Change in Quality of Life: Dyspnea
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the scales measure dyspnea.
  The range of score is 0-100; higher score = higher symptoms burden.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | -6.19 (4.88) | 7.12 (4.99)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.051, Mixed Models Analysis; Mean Difference (Net) = -13.31, Standard Error of Mean 6.62

15. Secondary Outcome: Change in Quality of Life: Insomnia
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the scales measure insomnia.
  The range of score is 0-100; higher score = better functioning.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 0.58 (6.37) | -3.49 (6.52)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.643, Mixed Models Analysis; Mean Difference (Net) = 4.07, Standard Error of Mean 8.71

16. Secondary Outcome: Change in Quality of Life: Appetite Loss
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the scales measure appetite loss The range of score is 0-100; higher score = higher symptoms burden.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | -4.16 (6.60) | 4.95 (6.73)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.290, Mixed Models Analysis; Mean Difference (Net) = -9.11, Standard Error of Mean 8.50

17. Secondary Outcome: Change in Quality of Life: Constipation
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the scales measure constipation.
  The range of score is 0-100; higher score = higher symptoms burden.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | -1.21 (4.02) | -11.19 (4.11)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.077, Mixed Models Analysis; Mean Difference (Net) = 9.99, Standard Error of Mean 5.49

18. Secondary Outcome: Change in Quality of Life: Diarrhea
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the scales measure diarrhea.
  The range of score is 0-100; higher score = higher symptoms burden.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 0.14 (3.32) | -5.13 (3.39)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.237, Mixed Models Analysis; Mean Difference (Net) = 5.27, Standard Error of Mean 4.38

19. Secondary Outcome: Change in Quality of Life: Financial Difficulties
Description: Assessed via self-report using the European Organization for the Research and Treatment of Cancer, Quality of Life Questionnaire (QLQ-C30, Version 3). The scale measures quality of life in 30 questions with 15 subscales. One of the scales measure financial difficulties.
  The range of score is 0-100; higher score = higher symptoms burden.
Time Frame: change from pre- to post-intervention (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 6.56 (4.54) | 5.41 (4.65)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.861, Mixed Models Analysis; Mean Difference (Net) = 1.15, Standard Error of Mean 6.49

20. Secondary Outcome: Moderate Aerobic Exercise
Description: The investigators will use the Physical Activity Questionnaire that measures this outcome in minutes.
Time Frame: baseline to 12 weeks
Population: A 12 week outcome was not available for one subject in the control group.
Measure: Mean (Standard Deviation); unit: Minutes of activity per week
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
Minutes of activity per week
  Baseline | 37.0 (46.4) | 58.8 (55.8)
  12 weeks: number analyzed (Participants) | 20 | 19
  12 weeks | 128.1 (212.4) | 75.3 (111.8)

21. Secondary Outcome: Vigorous Aerobic Exercise
Description: The investigators will use the Physical Activity Questionnaire that measures this outcome in minutes.
Time Frame: baseline to 12 weeks
Population: A 12 week outcome was not available for one subject in the control group.
Measure: Mean (Standard Deviation); unit: Minutes of activity per week
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
Minutes of activity per week
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  12 weeks: number analyzed (Participants) | 20 | 19
  12 weeks | 32.0 (82.5) | 17.4 (75.7)

22. Secondary Outcome: Change in C-reactive Protein (CRP)
Description: The investigators will obtain serum CRP, a marker of inflammation.
Time Frame: change from pre- to post-intervention (week 12)
Population: Only n=10 patients provided baseline and follow-up samples; 6 in the intervention group and 4 in the control group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 6 | 4
ng/mL | -1,381.34 (682.02) | -1,242.47 (918.90)

23. Secondary Outcome: Change in Leptin Level
Description: The investigators will obtain serum leptin, a marker of glucose control. .
Time Frame: change from pre- to post-intervention (week 12)
Population: Only n=10 patients provided baseline and follow-up samples; 6 in the intervention group and 4 in the control group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 6 | 4
ng/mL | 0.34 (3.28) | -3.31 (3.50)

24. Secondary Outcome: Change in Insulin Level
Description: The investigators will obtain serum insulin level, a measure of glucose control.
Time Frame: change from pre- to post-intervention (week 12)
Population: Only n=10 patients provided baseline and follow-up samples; 6 in the intervention group and 4 in the control group.
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 6 | 4
uIU/mL | 5.08 (7.29) | 8.32 (7.01)

25. Secondary Outcome: Programmed Death - Ligand
Description: The investigators will collect soluble PD- L1, a novel cancer marker.
Time Frame: change from pre- to post-intervention (week 12)
Population: Only n=10 patients provided baseline and follow-up samples; 6 in the intervention group and 4 in the control group.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 6 | 4
pg/mL | 1.22 (8.18) | -11.08 (11.17)

26. Secondary Outcome: Programmed Cell Death (PD-1)
Description: The investigators will collect soluble PD- 1, a novel cancer marker.
Time Frame: change from pre- to post-intervention (week 12)
Population: Only n=10 patients provided baseline and follow-up samples; 6 in the intervention group and 4 in the control group.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 6 | 4
pg/mL | 152.76 (45.51) | -67.03 (41.49)

ADVERSE EVENTS:
Time Frame: Twelve weeks.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20 | 1/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=20) | Control Group (N=20)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=20) | Control Group (N=20)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03352245/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03352245/ICF_001.pdf